CLINICAL TRIAL: NCT07277257
Title: Evaluating TRYPTYR as a Novel Therapy for Dry Eye in Patients With Sjögren's Syndrome
Brief Title: Evaluating a New Therapy for Dry Eye in Patients With Sjögren's Syndrome
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Center For Sight (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CFS25-004
Record Dates: First submitted 2025-12-02; First posted 2025-12-11 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Sjogren Syndrome With Keratoconjunctivitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study eye (Experimental): The study eye is the eye with the lower pre-drop unanesthetized Schirmer score performed at the baseline visit.
  Interventions: Drug: TRYPTYR (Acoltremon ophthalmic solution 0.003%)

INTERVENTIONS:
Drug: TRYPTYR (Acoltremon ophthalmic solution 0.003%) — Drop to be instilled before and after endpoint measurement.

SUMMARY:
This study will evaluate the effect of TRYPTYR in patients with Sjögren's syndrome-related dry eye disease. The goal is to determine whether TRYPTYR can improve symptoms and signs of dry eye in this specific patient population.

ELIGIBILITY:
Inclusion Criteria:

Subjects must fulfill the following conditions to qualify for enrollment into the trial

1. Adults over 18 years old with a diagnosis of dry eye disease (DED) secondary to Sjögren's Syndrome within the past 2 years.
2. History of using or desiring artificial tears for DED symptoms within the past 2 months.
3. Unanesthetized Schirmer's Test (UA ST) score ≥1 and < 10 mm/5 min and baseline total Corneal Fluorescein Staining (tCFS) score ≥2 and ≤ 15 (National Eye Institute, NEI, grading scale).

Exclusion Criteria:

Subjects with any of the following conditions on the eligibility exam may NOT be enrolled into the trial.

1. History of ocular surgery within the past 6 months.
2. Contact lens wear in either eye within 7 days of visit 1 (baseline) or use during study
3. On current topical treatment regimen for less than 3 months or anticipates any change to the regimen during the study period.
4. Use of topical steroid ocular medication or varenicline nasal spray within 4 weeks of baseline or during the study period.
5. Use of artificial tears within 2 hours prior to the baseline or study visit days.
6. Any known allergies to any component of the study drug.
7. Severe, uncontrolled autoimmune disease (e.g., rheumatoid arthritis, lupus). Uncontrolled is at the discretion of the PI. Subjects with severe systemic symptoms will not be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-12-02 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from pre-instillation to 3 minutes post-TRYPTYR instillation in study eye unanesthetized Schirmer's test at Visit 1 (baseline) | 3 minutes
  Unanesthetized Schirmer's test will be measured prior to instillation and then again 3 minutes after instillation of the TRYPTYR. The difference between the 2 measurements will be compared.

CONTACTS AND LOCATIONS:
Locations (1):
- Center For Sight, Venice, Florida, United States